CLINICAL TRIAL: NCT05387499
Title: A Phase 1, Randomised, Double-blind, Placebo-Controlled, Single Ascending Dose and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of NP-011 in Healthy Volunteers
Brief Title: A Study of NP-011 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nexel Co., Ltd. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP-011-001
Record Dates: First submitted 2022-05-04; First posted 2022-05-24 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-03

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Ascending Dose Phase (Experimental): Drug: NP-011 Dosage: 250μg, 500μg, 1000μg, 2000μg, 4000μg Dosage Form: Liquid for IV injection Route of Administration: Intravenous
  Interventions: Drug: NP-011 (Single Ascending Dose Phase)
- Multiple Ascending Dose Phase (Experimental): Drug: NP-011 Dosage: 1000μg, 2000μg, 4000μg Dosage Form: Liquid for IV injection Route of Administration: Intravenous
  Interventions: Drug: NP-011 (Multiple Ascending Dose Phase)
- Placebo (Placebo Comparator): Dosage Form: Liquid for IV injection Route of Administration: Intravenous
  Interventions: Other: NP-011 (Placebo)

INTERVENTIONS:
Drug: NP-011 (Single Ascending Dose Phase) — The participants will receive assigned single dose of NP-011 after a minimum 8 hour fast on Day 1
  Arms: Single Ascending Dose Phase
Drug: NP-011 (Multiple Ascending Dose Phase) — The participants will receive assigned dose of NP-011 after a minimum 8 hour fast once daily for 7 days
  Arms: Multiple Ascending Dose Phase
Other: NP-011 (Placebo) — The participants will receive single dose of NP-011 after a minimum 8 hour fast on Day 1 in Single Ascending Dose part and will receive once daily for 7 days after a minimum 8 hour fast in Multiple Ascending dose part of the study
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomised, double-blind, placebo-controlled, single ascending dose (SAD) and multiple ascending dose (MAD) study to evaluate the safety, tolerability, and pharmacokinetic of NP-011 in healthy volunteers.

DETAILED DESCRIPTION:
NP-011 is a truncated form of human MFG-E8 recombinant protein. NP-011 placebo has an identical formulation to the NP-011 drug product, prepared without the active pharmaceutical ingredient.

The study will be conducted in 2 parts:

Single Ascending Dose (SAD): The participants will be randomized to receive NP-011 (n= 6 per cohort) or placebo (n= 2 per cohort) on Day 1.

For all Part 1 cohorts, 2 sentinel participants will receive the first dose of IP (1 to receive NP-011, 1 to receive placebo) on Day 1. If dosing of the sentinel participants proceeds without clinically significant adverse events over 24 hours, the remaining participants in the cohort will be dosed at the discretion of the Principal Investigator (PI), according to the randomization schedule.

There are total five cohorts in Part 1 Cohort 1A: NP-011 250 μg or placebo (6:2) Cohort 1B: NP-011 500 μg or placebo (6:2) Cohort 1C: NP-011 1000 μg or placebo (6:2) Cohort 1D: NP-011 2000 μg or placebo (6:2) Cohort 1E: NP-011 4000 μg or placebo (6:2)

Multiple Ascending Dose (MAD): The part 2 progress after the completion of Day 8 assessments in Cohort 1E upon satisfactory review of all available safety data by the SMC.

Participants will be enrolled into 3 sequential cohorts in Part 2. Dose levels for Part 2 cohorts may be revised by agreement with the SMC and based on emerging safety and PK data.

Cohort 2A: NP-011 1000 μg or placebo (6:2) Cohort 2B: NP-011 2000 μg or placebo (6:2) Cohort 2C: NP-011 4000 μg or placebo (6:2)

The participants will be randomized to receive the NP-011 (n= 6 per cohort) or placebo (n=2 per cohort)

The safety and pharmacokinetic data will be reviewed by SMC in both the parts (SAD and MAD) prior to the decision to increase or decrease the dose level for the next cohort or expand the number of participants in a cohort (to a maximum of an additional 8 participants at a given dose level).

ELIGIBILITY:
Inclusion Criteria:

1. Normal healthy volunteers with an age of 18 to 65 years inclusive at the time of informed consent.
2. Participants can be of any ethnicity or race, excluding Asian by self-declaration. For the purposes of this protocol, Asian is defined as a person having origins in any of the original peoples of the Far East, Southeast Asia, or the Indian subcontinent, including for example, Cambodia, China, India, Japan, Korea, Malaysia, Pakistan, Philippines, Thailand, and Vietnam. If an individual identifies as mixed race, exclusion will occur if the proportion of self-declaration as Asian exceeds 25%.
3. Participants must be in good general health, in the opinion of the Investigator, with no significant medical history (ie, history of childhood asthma [resolved] is acceptable; history of depression [non-hospitalised, medicated] or migraines is not acceptable), and no clinically significant abnormalities on physical examination at Screening and/or before administration of the initial dose of IP.
4. Participants must have documented evidence of receipt of licensed COVID-19 vaccinations as per the current Australian Technical Advisory Group on Immunisation (ATAGI) guidelines and be fully vaccinated as per local guidelines.
5. Participants must have a BMI between > 18.0 and < 32.0 kg/m2 at Screening.
6. Participants must have clinical laboratory values within normal range as specified by the testing laboratory, unless deemed not clinically significant by the Investigator or delegate. A single repeat test can be performed for clinically significant abnormal values, at the discretion of the Investigator.
7. Participants must be a non-smoker and must not have used any tobacco products within 2 months prior to Screening, or if a smoker, they must smoke no more than 2 cigarettes or equivalent per week.
8. Participants must have no relevant dietary restrictions (restrictions that would prevent consumption of the standard meals to be provided), and be willing to consume standard meals provided.
9. Females must be non-pregnant and non-lactating, and must use an acceptable, highly effective double contraception from Screening until 30 days after last dose of IP, including the follow-up period. Double contraception is defined as a condom AND one other form of the following:

   * Established hormonal contraception (with approved oral contraceptive pills [OCPs], long-acting implantable hormones, injectable hormones);
   * A vaginal ring or an intrauterine device (IUD);
   * Documented evidence of surgical sterilisation at least 6 months prior to Screening (eg, tubal occlusion, hysterectomy, bilateral salpingectomy, or bilateral oophorectomy for women or vasectomy for men, provided the male partner is a sole partner).

   Women not of childbearing potential must be post-menopausal for ≥ 12 months. Post-menopausal status will be confirmed through testing of follicle-stimulating hormone (FSH) levels ≥ 40 IU/L at Screening for amenorrhoeic female participants. Females who are abstinent from heterosexual intercourse will also be eligible.

   Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not considered highly effective methods of birth control. Participant complete abstinence for the duration of the study and for 1 month after the last study treatment is acceptable.

   Female participants who are in exclusively same-sex relationships are not required to use contraception.

   Woman of childbearing potential (WOCBP) must have a negative pregnancy test at Screening and Day 1 and be willing to have additional pregnancy tests as required throughout the study.

   Males must be surgically sterile (> 30 days since vasectomy with no viable sperm), abstinent, or if engaged in sexual relations with a WOCBP, the participant and his partner must be surgically sterile (eg, tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or using an acceptable, highly effective contraceptive method from Screening until study completion, including the follow-up period, and for at least 90 days post final dose. Acceptable methods of contraception include the use of condoms and the use of an effective contraceptive for the female partner that includes: OCPs, long-acting implantable hormones, injectable hormones, a vaginal ring, or an IUD. Participants with same-sex partners (abstinence from penile-vaginal intercourse) are eligible when this is their preferred and usual lifestyle.
10. Male participants must not donate sperm for at least 90 days after the last dose of IP, and female participants must not donate ovum for at least 30 days after the last dose of IP.

Exclusion Criteria:

1. Use of any IP or investigational medicinal device within 30 days prior to treatment, or 5 half-lives of the product, whichever is the longest.
2. Prior or ongoing medical conditions, medical history, physical findings, or laboratory abnormality that, in the Investigator's opinion, could adversely affect the safety of the participant or confound treatment assessment.
3. Allergy or hypersensitivity to the IP or any of its constituents.
4. History of allergic or anaphylactic reactions that are considered severe in the opinion of the Investigator (with the allowance of well-managed allergies such as allergic rhinitis, eczema, stinging insect allergies, and pollen allergies).
5. Any history of cardiac disease.
6. Abnormal ECG findings at Screening that are considered by the Investigator to be clinically significant.
7. Use of or anticipated use of any prescription drugs (other than hormonal contraception; OCPs, long-acting implantable hormones, injectable hormones, a vaginal ring, or an IUD), over-the-counter (OTC) medication, herbal remedies, supplements, or vitamins 2 weeks prior to dosing and during course of study without prior approval of the Investigator and MM. Simple analgesics (paracetamol, nonsteroidal anti-inflammatory drugs [NSAIDs]) are permitted at 1 or 2 therapeutic doses per week at the discretion of the Investigator.
8. Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including the follow-up period.
9. Presence of any underlying physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the participant will comply with the protocol or complete the study per protocol.
10. Blood donation or significant blood loss within 60 days prior to the first IP administration.
11. Plasma donation within 7 days prior to the first IP administration.
12. Fever (body temperature > 38°C) or symptomatic viral or bacterial infection within 2 weeks prior to Screening.
13. History of malignancy, except for non-melanoma skin cancer, excised more than 2 years ago and cervical intraepithelial neoplasia that has been successfully cured more than 5 years prior to Screening.
14. History or presence of a condition associated with significant immunosuppression (significant in the opinion of the Investigator).
15. History of life-threatening infection (eg, meningitis).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of single and multiple doses of NP-011 through the incidence, nature and severity of adverse events | Screening to end of the follow up period; up to 36 and 56 days for Single Ascending Dose and Multiple Ascending Dose
  Adverse Events will be coded using the most current version of the MedDRA®

SECONDARY OUTCOMES:
To characterize the plasma pharmacokinetics (PK) of NP-011 in healthy volunteers | Screening to end of the follow up period; up to 36 and 56 days for Single Ascending Dose and Multiple Ascending Dose
  Parameter: maximum concentration (Cmax)
To characterize the plasma pharmacokinetics (PK) of NP-011 in healthy volunteers | Screening to end of the follow up period; up to 36 and 56 days for Single Ascending Dose and Multiple Ascending Dose
  Parameter: time to maximum concentration (Tmax)
To characterize the plasma pharmacokinetics (PK) of NP-011 in healthy volunteers | Screening to end of the follow up period; up to 36 and 56 days for Single Ascending Dose and Multiple Ascending Dose
  Parameter: area under the concentration-time curve (AUC)
To characterize the immunogenicity of NP-011 in healthy volunteers by assessing the development of anti-drug-antibodies (ADA) through change from baseline in neutralizing antibody titers for NP-011 after single and multiple doses. | Screening to end of the follow up period; up to 36 and 56 days for Single Ascending Dose and Multiple Ascending Dose

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Gehlert, Principal Investigator — CMAX Clinical Research Pty Ltd
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No